CLINICAL TRIAL: NCT06919757
Title: Early Lung Function Trajectories: Comparison Between Infants With Intrauterine Growth Restriction and Appropriately Grown Ones.
Brief Title: Early Lung Function Trajectories: Comparison Between Infants With and Without Intrauterine Growth Restriction.
Acronym: ELFIGO
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6642
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Intrauterine Growth Retardation (IUGR); Lung Function Tests; Preterm Infant; Respiratory Monitoring
Keywords: lung volume measurements; pulmonary function test; preterm birth; intrauterine growth retardation; oxygen saturation/physiology
MeSH Terms: conditions — Fetal Growth Retardation; Premature Birth | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants born preterm with history of IUGR: preterm infants with history of intrauterine growth restriction
  Interventions: Diagnostic Test: fetal ultrasound to assess lungs, heart and diaphragm
- Infants born preterm without history of IUGR: preterm infants without history of intrauterine growth restriction
  Interventions: Diagnostic Test: fetal ultrasound to assess lungs, heart and diaphragm

INTERVENTIONS:
Diagnostic Test: fetal ultrasound to assess lungs, heart and diaphragm — The potential association between fetal ultrasound parameters (estimation of lung volumes, diaphragmatic thickness and contractility, cardiac thickness and kinetics), perinatal complications and respiratory function in the first years of life will be studied. Variables include: neonatal complications, non-invasive markers of respiratory status during neonatal admission (e.g. peripheral oxygen saturation/rfaction of inspired oxygen ratio among others), lung function tests in the first two years of life.
  Other Names: lung function tests

SUMMARY:
During intrauterine life, some babies are smaller or grow less than expected. This fetal growth abnormality, called fetal growth restriction (FGR), can be diagnosed by ultrasound. Since there are currently no curative treatments for this condition, nor methods to optimize the growth of babies in the womb, the only effective strategy is intensive monitoring of fetal conditions, accompanied by early planning of delivery.

The diagnosis of early FGR (i.e. diagnosed before 32 weeks of gestation) confers a greater risk of short- and long-term respiratory problems.

The study aims to examine the association between parameters that can be assessed during pregnancy by ultrasound, such as the estimate of lung volumes, the thickness and contractility of the diaphragm, and cardiac kinetics, and any perinatal complications and respiratory function in the first years of life of premature infants, both with and without evidence of fetal growth pathology. Therefore, the study is divided into two phases: a prenatal and a postnatal phase.

The study includes two groups of patients:

1. Study group: Fetuses and preterm infants with a prenatal history of FGR;
2. Control group: Preterm infants without a prenatal history of FGR followed during neonatal follow-up.

Pregnant women with fetuses with FGR are followed at the Ultrasound clinics dedicated to Growth Pathology.

These pregnancies usually receive weekly ultrasound monitoring, which includes a Doppler study of the maternal and fetal circulation and an estimate of fetal weight every two weeks. Cardiotocographic monitoring is also planned once or twice a week, depending on fetal well-being.

The child will be assessed from a respiratory point of view during hospitalization and subsequently in the outpatient clinic, as required by clinical practice.

He/she will undergo respiratory function tests. Visits are scheduled at 3, 6, 12 and 24 months of corrected age, during which at least two respiratory function tests will be performed.

In addition, routine clinical data (personal data, medical history, blood tests, biological and instrumental tests) present in the medical record of the child will be collected.

Data from preterm infants without fetal growth restriction will be collected after informed consent. These infants are routinely followed at our Institution and undergo clinical assessment and lung function tests in the first two years of life as previously indicated.

ELIGIBILITY:
Inclusion Criteria:

* Fetuses and Infants born before 32 weeks of gestation, with and without fetal growth restriction

Exclusion Criteria:

* Lack of informed consent
* Need for palliative care
* Major malformations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fetuses and Infants born before 32 weeks of gestation, with and without fetal growth restriction
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Bronchopulmonary dysplasia | 36 weeks post-menstrual age
  Respiratory support at 36 weeks post-menstrual age
Death | 2 years of life
  occurrence of death during NICU admission or afterwards
Lung function data | 2 years of life
  Data from the Tidal breathing flow volume test and multiple breath nitrogen washout

SECONDARY OUTCOMES:
Peripheral oxygen saturation/fraction on inspired oxygen ratio (SFR) | 16 weeks of life
  non-invasive ratio between peripheral oxygen saturation/fraction on inspired oxygen ratio
Peripheral oxygen saturation/fraction on inspired oxygen ratio divided by mean airway pressure (SFR/P) | 16 weeks of life
  non-invasive ratio between peripheral oxygen saturation/fraction on inspired oxygen ratio and mean airway pressure

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nobile, MD, PhD, MSc, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nobile S, Marchionni P, Carnielli VP. Neonatal outcome of small for gestational age preterm infants. Eur J Pediatr. 2017 Aug;176(8):1083-1088. doi: 10.1007/s00431-017-2957-1. Epub 2017 Jun 28. PMID 28660312
- [Background] Jensen EA, Foglia EE, Dysart KC, Simmons RA, Aghai ZH, Cook A, Greenspan JS, DeMauro SB. Adverse effects of small for gestational age differ by gestational week among very preterm infants. Arch Dis Child Fetal Neonatal Ed. 2019 Mar;104(2):F192-F198. doi: 10.1136/archdischild-2017-314171. Epub 2018 May 5. PMID 29730594
- [Background] D'Agostin M, Di Sipio Morgia C, Vento G, Nobile S. Long-term implications of fetal growth restriction. World J Clin Cases. 2023 May 6;11(13):2855-2863. doi: 10.12998/wjcc.v11.i13.2855. PMID 37215406
- [Background] Arigliani M, Stocco C, Valentini E, De Pieri C, Castriotta L, Ferrari ME, Canciani C, Driul L, Orsaria M, Cattarossi L, Cogo P. Lung function between 8 and 15 years of age in very preterm infants with fetal growth restriction. Pediatr Res. 2021 Sep;90(3):657-663. doi: 10.1038/s41390-020-01299-0. Epub 2021 Jan 19. PMID 33469172
- [Background] Nobile S, Marchionni P, Gidiucci C, Correani A, Palazzi ML, Spagnoli C, Rondina C; Marche Neonatal Network; Carnielli VP. Oxygen saturation/FIO2 ratio at 36 weeks' PMA in 1005 preterm infants: Effect of gestational age and early respiratory disease patterns. Pediatr Pulmonol. 2019 May;54(5):637-643. doi: 10.1002/ppul.24265. Epub 2019 Jan 27. PMID 30688034
- [Background] Salem Y, Willers CC, Amylidi-Mohr S, Kentgens AC, Stranzinger E, Latzin P, Raio L, Yammine S. Low Birth Weight and Impaired Later Lung Function: Results from a Monochorionic Twin Study. Ann Am Thorac Soc. 2022 Nov;19(11):1856-1864. doi: 10.1513/AnnalsATS.202112-1349OC. PMID 35580242